CLINICAL TRIAL: NCT05629117
Title: The Effects of Personalized Diabetes Text Messaging (DB-TEXT) Combined With Peer Support Education in Patients With Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Personalized Diabetes Text Messaging (DB-TEXT) Combined With Peer Support Education in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No.1738/UN25.8/KEPK/DL/2022
Record Dates: First submitted 2022-11-11; First posted 2022-11-29 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes Text Messaging (DB-TEXT), peer support education, type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Diabetes Text Messaging (DB-TEXT) combined with Peer Support Education Group (Experimental): Patients who are assigned to the DB-TEXT+PSE group will receive personalized short text message services twice weekly at approximately noon on Monday and Thursday for three months (12 weeks). Additionally they will receive peer support education weekly during three month.
  Interventions: Behavioral: Personalized Diabetes Text Messaging (DB-TEXT) combined with Peer Support Education
- Personalized Diabetes Text Messaging (DB-TEXT) Group (Active Comparator): The participants in the Personalized DB-TEXT group will receive the personalized short text message twice weekly at approximately noon on Monday and Thursday for three months (12 weeks).
  Interventions: Behavioral: Personalized Diabetes Text Messaging (DB-TEXT)
- Control Group (No Intervention): Health education related to diabetes management will be provided to the control group once a month during three months

INTERVENTIONS:
Behavioral: Personalized Diabetes Text Messaging (DB-TEXT) combined with Peer Support Education — Patients who are assigned to the DB-TEXT+PSE group will receive personalized short text message services twice weekly at approximately noon on Monday and Thursday for three months (12 weeks). Furthermore, they will receive the peer support education weekly from the peer supporter by telephone during three months
  Arms: Personalized Diabetes Text Messaging (DB-TEXT) combined with Peer Support Education Group
Behavioral: Personalized Diabetes Text Messaging (DB-TEXT) — Personalized Diabetes Text Messaging (DB-TEXT)
  Arms: Personalized Diabetes Text Messaging (DB-TEXT) Group

SUMMARY:
The purpose of this study to investigate the effects of personalized diabetes text messaging (DB-TEXT) combined with PSE in patients with type 2 diabetes. This study is an assessor-blinded, three-arm, parallel randomized controlled trial. Additionally, the investigators will use the CONSORT guidelines to report of trial finding. A diabetes management centers in East Java Province will be recruited for the participants from December 2022 to March 2023. The investigators will include participants who had been diagnosed with poorly controlled type 2 diabetes (having HbA1C level of > 7% in the past three months), and who were 17 years or older (the legal age to provide informed consent in Indonesia) and having their own mobile phone. People who could not read or write Indonesian; had medical diagnostic with cognitive impairments, psychiatric disorders, or were diagnosed with cancer before the study will be excluded from the study. The outcomes of the study including demographic and disease characteristic, clinical outcomes, fatigue, sleep quality, depression, and quality of life. For the clinical outcomes, will be measured in laboratory test in diabetes management centers. Fatigue level will be measured using the Multidimensional Fatigue Inventory-20 (MFI-20), sleep quality will be measured using a Pittsburgh Sleep Quality Index (PSQI), the Beck Depression Inventory-Second Edition (BDI-II) will be used to measure the depression level, and the Diabetes Quality of Life-Brief Clinical Inventory (The DQoL-BCI) will be used to assess the quality of life.

DETAILED DESCRIPTION:
Background :

Our early component network meta-analysis (CNMA) study showed that short message service (SMS) and peer support education (PSE) are the most effective component of digitally assisted intervention in improving HbA1C level in type 2 diabetes.

Purposes:

The purpose of this study to investigate the effects of personalized diabetes text messaging (DB-TEXT) combined with PSE in patients with type 2 diabetes.

Methods:

This study is an assessor-blinded, three-arm, parallel randomized controlled trial (RCT). Additionally, the investigators will use the CONSORT guidelines to report of trial finding. A diabetes management centers in East Java Province will be recruited for the participants from December 2022 to March 2023. The investigators will include participants who had been diagnosed with poorly controlled type 2 diabetes (having HbA1C level of > 7% in the past three months), and who were 17 years or older (the legal age to provide informed consent in Indonesia) and having their own mobile phone. People who could not read or write Indonesian; had medical diagnostic with cognitive impairments, psychiatric disorders, or were diagnosed with cancer before the study will be excluded from the study.The outcomes of the study including demographic and disease characteristic, clinical outcomes, fatigue, sleep quality, depression, and quality of life. For the clinical outcomes, will be measured in laboratory test in diabetes management centers. Fatigue level will be measured using the Multidimensional Fatigue Inventory-20 (MFI-20), sleep quality will be measured using a Pittsburgh Sleep Quality Index (PSQI), the Beck Depression Inventory-Second Edition (BDI-II) will be used to measure the depression level, and the Diabetes Quality of Life-Brief Clinical Inventory (The DQoL-BCI) will be used to assess the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants who had been diagnosed with poorly controlled type 2 diabetes (having HbA1C level of > 7% in the past three months)
* Participants ho were 17 years or older (the legal age to provide informed consent in Indonesia)
* having their own mobile phone

Exclusion Criteria:

* People who could not read or write Indonesian
* Had medical diagnostic with cognitive impairments
* Psychiatric disorders, or were diagnosed with cancer

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1C level | at baseline, 3 months, 6 months
  HbA1C level of participants will be assessed in the laboratory test in hospital
Changes in fasting blood glucose level | at baseline, 3 months, 6 months
  Fasting blood glucose level of participants will be assessed using glucometer
Changes in Lipids level including total cholesterol, Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL) , and triglycerides | at baseline, 3 months, 6 months
  The total cholesterol, LDL, HDL, and triglycerides of the participants will assessed in the laboratory test in hospital
Changes in Blood Pressure Level including Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) | at baseline, 3 months, 6 months
  Blood pressure of participants will be measured using sphygmomanometer

SECONDARY OUTCOMES:
Changes in Fatigue | At baseline, 3 months, 6 months
  Fatigue levels of participants will be assessed using a Multidimensional Fatigue Inventory-20 (MFI-20). MFI-20 contains 20 items and five subscales, general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue.
Changes in Sleep Quality | At baseline, 3 months, 6 months
  Sleep quality of the participants will be measured using The Pittsburgh Sleep Quality Index (PSQI). PSQI assesses self-reported sleep quality and sleep disturbance in the preceding month.
Changes in Depression | At baseline, 3 months, 6 months
  The depression levels of participants will be assessed using the Beck Depression Inventory-Second Edition (BDI-II). There are 21 items on the BDI-II that measure subjective depression symptoms over the preceding 2 weeks
Changes in Quality of Life | At baseline, 3 months, 6 months
  Quality of life of the participants will be measured using the Diabetes Quality of Life-Brief Clinical Inventory (The DQoL-BCI). DQoL-BCI contains 15 questions. Using a Likert scale of 5 points, participants can assess their satisfaction with each DQoL-BCI item (1=Very Dissatisfied/All the Time, 2=Moderately Dissatisfied/Sometimes, 3=Neither/Sometimes, and 4=Moderately Satisfied/Very Seldom).

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Xinyi District, Taiwan

IPD SHARING:
Plan to Share IPD: No